CLINICAL TRIAL: NCT04757402
Title: Role of Preoperative Counselling With NSQIP Surgical Risk Calculator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Bikash Khadka, Anesthesiologist, Nepal Mediciti Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2077/0019
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Satisfaction, Patient
Keywords: NSQIP Surgical risk calculator; Preoperative counselling; Anxiety
MeSH Terms: conditions — Patient Satisfaction; Anxiety Disorders | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): All eligible candidates will be receiving standard preoperative counselling as per the hospital standards and protocols. The patient will fill five-points Amsterdam Preoperative Anxiety and Information Scale (APAIS) form for anxiety evaluation and Seven-points Likert Scale form for satisfaction regarding the counselling.
  Interventions: Other: Counselling with NSQIP Surgical risk calculator
- NSQIP Arm (Experimental): All eligible candidates will be receiving standard preoperative counselling as per the control arm PLUS the risk will be explained using the scores from the NSQIP surgical risk calculator. The anxiety and the satisfaction scores will be recorded as in the control arm.
  Interventions: Other: Counselling with NSQIP Surgical risk calculator

INTERVENTIONS:
Other: Counselling with NSQIP Surgical risk calculator — Use of NSQIP surgical risk calculator to check for patient satisfaction regarding pre operative counseling.

SUMMARY:
Surgical patients undergo preoperative counseling which varies in quality and duration. Proper communication during the preoperative consultation can deliver relevant health information and guide improvement of perioperative health status. The methods, however, are non-standardized and the explanation of the postoperative course is generally vague or varies from person to person. We hypothesize that high-risk patients who receive pre-operative counseling with the help of the NSQIP surgical risk calculator compared to the current standard of care will have higher satisfaction concerning information on the perioperative journey.

DETAILED DESCRIPTION:
The control arm will receive standard preoperative counselling and written consent will be taken.

The NSQIP arm will receive standard preoperative counselling along with the details provided by NSQIP Surgical risk calculator and written consent will be taken.

Anxiety among the patients will be accessed with the use of Preoperative anxiety measured by Amsterdam Preoperative Anxiety and Information Scale (APAIS) questionnaire written in Nepali.

Duration of counselling period will be noted from the start of counselling session till the consent is signed.

ELIGIBILITY:
Inclusion Criteria:

* ASA III or above and/or age above 65 high-risk surgical patients undergoing surgery at Nepal Mediciti Hospital

Exclusion Criteria:

* Adults who cannot consent Pregnant women Non-Nepali speakers Consent by surrogate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
The difference in patient satisfaction as assessed by a 7-point Likert scale | 5 MONTHS
  The study will compare patient satisfaction scores between the two arms of the study groups to determine if there is a difference in patient satisfaction. It will be based on a scale of 1 to 7, 7 being the most satisfied and 1 being the least.

SECONDARY OUTCOMES:
Preoperative anxiety measured by Amsterdam Preoperative Anxiety and Information Scale (APAIS) questionnaire written in Nepalese | 5 months
  Anxiety evaluation during preoperative counselling will be done by APAIS using a five point scale,5 being the most anxious and 1 being the least.
Duration of counseling | 5 months
  time taken to complete preoperative counseling which will be noted from start of counseling to the time when consent is signed.

CONTACTS AND LOCATIONS:
Overall Officials: Apurb Sharma, MD, Study Chair — Nepal Mediciti Hospital
Locations (1):
- Bikash Khadka, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 10 months
Access Criteria: an email with explanations for the need of data

REFERENCES:
- [Background] Sigdel S, Ozaki A, Basnet M, Kobashi Y, Pradhan B, Higuchi A, Uprety A. Anxiety evaluation in Nepalese adult patients awaiting cardiac surgery: A prospective observational study. Medicine (Baltimore). 2020 Feb;99(9):e19302. doi: 10.1097/MD.0000000000019302. PMID 32118748